CLINICAL TRIAL: NCT02734459
Title: A Multi Center, Open Label, Randomized, Two- Treatment, Single Dose, Crossover, Bioequivalence Study To Compare The Pharmacokinetics Of Marketed Product TobraDex® (Tobramycin And Dexamethasone Ophthalmic Ointment) To An Experimental Ophthalmic Sterile Ointment Containing Tobramycin 0.3% And Dexamethasone 0.1% W/W In Aqueous Humor In Patients Undergoing Indicated Cataract Surgery
Brief Title: A Bioequivalence Study to Compare the Pharmacokinetics (PK) Of Marketed Product TobraDex® To An Experimental Ophthalmic Sterile Ointment Containing Tobramycin And Dexamethasone In Aqueous Humor In Patients Undergoing Indicated Cataract Surgery
Acronym: TBO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Semler Research Center Pvt. Ltd. (Industry)
Collaborators: Genzum Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: S-10-084
Record Dates: First submitted 2016-03-24; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Bilateral Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tobramycin and dexamethasone ophthalmic test ointment (Experimental): The test drug (tobramycin is an aminoglycoside antibiotic and dexamethasone is a corticosteroid) will be administered in one eye before the cataract surgery.
  Interventions: Drug: cataract surgery
- TobraDex® ointment (Active Comparator): The reference drug (tobramycin is an aminoglycoside antibiotic and dexamethasone is a corticosteroid) will be administered in another eye before the cataract surgery.
  Interventions: Drug: cataract surgery

INTERVENTIONS:
Drug: cataract surgery — the patient will be dosed with the study drug into the "V" pocket is formed between the eye ball and the lower eyelid during cataract surgery.

SUMMARY:
Each patient will be randomized to receive one dose of the test article in one eye and one dose of the reference formulations in the contralateral eye. One eye will be selected as the initial eye for cataract surgery and aqueous humor collection and hence will be dosed and operated on first. Followed by the second eye which will be dosed no early than a week followed by aqueous humor collection as per specified time points and no later than 35 days following the first eye again prior to the cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female 18 years of age and above
* Presence of visually significant cataracts in both eyes
* Have a chief complaint consistent with visually significant cataracts
* Be able to communicate effectively with the study personnel and be able to understand and follow directions
* Be medically fit with clinically acceptable laboratory profiles and ECG
* Be willing to carry out the required pre op directions and post op care and be able to make the scheduled appointment
* Have given the written informed consent for participation in the study
* In addition, female patients of child bearing potential age must have a negative urine pregnancy test

Exclusion Criteria:

* Participation in any ophthalmic indicative bioavailability/ bioequivalence/ Pharmacokinetic study or received an ophthalmic indicative investigational drug within a period of three months prior to screening
* Presence or history of recent viral corneal disorder or active corneal condition which is contraindicated.
* Presence or history of uveitis or uveitis
* Presence of retinal disorders
* Ocular trauma within three months of the trial
* Patients who had received topical and or systemic/ oral steroids
* Uncontrolled diabetes
* History of any allergies
* Known hypersensitivity or allergy to TobraDex® in combination or its components
* Clinical laboratory test values outside the acceptable reference range and when confirmed on re-examination deemed to be clinically significant as determined by the investigator(s)
* Clinically significant illness during 3 weeks prior to Visit 1 (as determined by the investigators)
* Presence of a clinically significant systemic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Concentration of dexamethasone in aqueous humor at different time points after administration of a single dose of each of the two drugs. | 30 min - 8 hours
  A series of aqueous humor samples will be collected from each eye of each patient.

OTHER OUTCOMES:
Time at which maximum mean drug concentration (Tmax) is achieved, in aqueous humor after the administration of test and reference drugs. | 30 min - 8 hours
AUC under the concentration-time curve from time-zero to the time t for test and reference drugs | 30 min - 8 hours
Maximum drug concentration (Cmax) achieved, in aqueous humor after the administration of test and reference drugs. | 30 min - 8 hours